CLINICAL TRIAL: NCT04124588
Title: A Prospective, Multicenter, Randomized Controlled Trial to Evaluate Safety and Effectiveness of Endoscopic Hemostactic Powder, 'Nexpowder' for Hemostatic Treatments of Nonvariceal, Upper Gastrointestinal Bleeding
Brief Title: Effectiveness of 'Nexpowder' for Hemostatic Treatments of Nonvariceal, Upper Gastrointestinal Bleeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Next Biomedical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NEXTBIO-632-EWD3
Record Dates: First submitted 2019-10-09; First posted 2019-10-11 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Nonvariceal Upper Gastrointestinal Bleeding

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): "After" achieving initial hemostasis only with the standard-of-care, endoscopic hemostatic therapie(s)
  Interventions: Device: Nexpowder (Hemostatic powder); Device: Conventional Technique
- Control gruop (Active Comparator): "After" achieving initial hemostasis only with the standard-of-care, Wrap up the first endoscopy without adding an additional procedure.
  Interventions: Device: Conventional Technique

INTERVENTIONS:
Device: Nexpowder (Hemostatic powder) — Nexpowder generates gelation-effects when the powder comes into contact with water, forms a physical barrier to control hemorrhage, preserve ulcer sites and thereby demonstrates its effective hemostatic performance. Hydrogels, which turned into gel-formation through water contacts in the gastrointestinal tract protect the wound sites for over 24 hours, are subsequently detached from the lesion, and completely excreted from the patient body system within 3 days.
  Arms: Test group
Device: Conventional Technique — Argon Plasma Coagulation, Coagulation including Forcep, Hemoclipping, Band Ligation, Epinephrine or Absolute Alcohol Injecction can be used as standard-of-care hemostatic treatment(s).

SUMMARY:
A prospective, multi-center, randomized controlled trial to evaluate safety and effectiveness of endoscopic hemostatic powder, 'Nexpowder' for hemostatic treatments of nonvariceal upper gastrointestinal bleeding.

This study is a prospective, multi-center, single blind (for patients), controlled investigation planned to evaluate safety and effectiveness of Nexpowder with 352 subject patients.

DETAILED DESCRIPTION:
This investigational study is designed to compare effectiveness of using the standard-of-care hemostatic therapy only, versus the standard-of-care hemostatic therapy plus an additional hemostatic treatment using Nexpower for patients with nonvariceal, upper gastrointestinal bleeding from ulcers with high-risk stigmata (Forrest classification Ia, Ib, or IIa).

The primary end-points will be evaluated by assessing the rates of re-bleeding, which occur over three (3) days following initial hemostasis achieved with the standard-of-care hemostatic therapy.

Secondary end-points consist of evaluating three items: 1) Ease of use of Nexpowder applied for the test group after reaching initial hemostasis, 2) Nexpowder device malfunction and 3) safety follow-up to check occurrence of adverse event(s)/re-bleeding at 30-day (+5) time point.

Only the subjects whose initial hemostasis has been achieved will be registered for this investigation but those who initial hemostasis has failed to be reached with the standard-of-care therapie(s) shall not be registered for this investigation.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female with age of older than 19 years.
* Patients showing non-variceal upper GI bleeding symptoms
* An endoscopic examination indicates that the patients's ulcer is categorized Class Ia, Ib, or IIa according to the Forrest Classifications.

Exclusion Criteria:

* Pregnant or breast-feeding patients

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-10-12 (Actual); Study Completion 2021-11-11 (Actual)

PRIMARY OUTCOMES:
The rates of re-bleeding | 3 days
  Assessing the rates of re-bleeding, which occur over three (3) days following initial hemostasis achieved with the standard-of-care hemostatic therapy.

SECONDARY OUTCOMES:
Incidence of Treatment-Adverse Events & Long term Re-bleeding | 30 days (+5)
  Safety follow-up to check occurrence of adverse event(s)/re-bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Eunhye Lee, Ph.D, Study Director — NEXTBIOMEDICAL CO., LTD.
Locations (3):
- South Korea (3):
  - Soon Chun Hyang University Bucheon Hospital, Gyeonggi-do
  - Gachon Gil Hospital, Incheon
  - Inha University Hospital, Incheon

REFERENCES:
- [Derived] Shin J, Cha B, Hong J, Kwon KS, Lee E, Maeng JH, Chung JW, Park DK, Kim YJ, Kwon KA, Kim JH, Seo KS, Hong SJ, Kim KO. Prevention of rebleeding after primary haemostasis using haemostatic powder in non-variceal upper gastrointestinal bleeding: a multicentre randomised controlled trial. Gut. 2025 Oct 8;74(11):1821-1827. doi: 10.1136/gutjnl-2024-332459. PMID 40360231